CLINICAL TRIAL: NCT05964712
Title: Effects of Therapies in the Acromegaly Disease: Acral Morpho-functional Study
Acronym: ACROMORFO
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: Politecnico di Milano (Other)
Responsible Party: Sponsor
Other Study IDs: 40C901
Record Dates: First submitted 2023-03-02; First posted 2023-07-28 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum dosage of GH and IGF-1
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Population # 1: De novo patients with acromegaly, diagnosed according to Endocrine Society guidelines, aged equal or above 18 years old
  Interventions: Procedure: Medical surgery therapy
- Population # 2: Acromegalic patients with different disease status (active disease despite ongoing therapies, controlled disease under medical therapy, and disease remission), aged equal or above 18 years old

INTERVENTIONS:
Procedure: Medical surgery therapy — De novo patients with acromegaly will undergo medical/surgical therapy of this disease, according to the guidelines of the Endocrine Society. In this population (group #1) morpho-functional examinations together with the evaluation of the stage of the disease, with serum dosage of GH and IGF-1, will be performed at baseline and at months 3, 6 and 12 after initiating the treatment.
  Groups: Population # 1

SUMMARY:
Acromegaly is a rare chronic disease due to excessive secretion of growth hormone (GH) and insulin-like growth factor-I (IGF-I), caused in over 98% of cases by GH-secreting pituitary adenoma. Prolonged exposure to GH/IGF-I excess is the cause of increased mortality and morbidity in these patients. Arthropathy occurs in about 75% of acromegalic patients. Any joint may be affected, with the development of osteoarthritis, arthralgia, and an increase in fracture risk.

The aims of the present project are to evaluate the dimensions of hands and feet with the 3D scanner method and to perform a quantitative analysis of movement through Gait Analysis technique in de novo patients with acromegaly (group # 1) and in patients with different disease status (group #2).

DETAILED DESCRIPTION:
This is an observational, prospective study that aims to evaluate the effect of acromegalic disease and medical/surgical therapy on acral morpho-functional alterations.

To outline the morphological characteristics of the extremities (hands and feet), a three-dimensional laser scanning system will be used able to measure the geometrical and volumetric characteristics of the hands and feet of these subjects. The three-dimensional scanning system that will be used is the portable FastScan system (marketed by Rodin), previously used for the volumetric evaluation of the lower and upper limbs of subjects suffering from lymphedema and lipedema. The processing of the image and the parameters will be carried out through two softwares: Rodin4DScan, which carries out the reconstruction of the shape after the scan, and Rodin4D, which allows the construction of the final shape and allows the processing of the various parameters to the morphology of the extremity.

The following tests will be used to characterize posture and balance control during walking:

* maintenance of the bipedal indifferent orthostatic posture, with open and closed eyes;
* walking on level ground, barefoot, at natural speed (10 m walking test)

The instrumentation (BTS GAITLAB) that will be used consists of:

* 8-camera stereophotogrammetric system (SMART DX, BTS-Bioengineering, IT);
* two dynamometric platforms (AMTI, USA);
* a baropodometric platform (P-WALK; BTS-Bioengineering, IT).

The variables analyzed will be divided according to the administered tests:

1. maintenance of the orthostatic posture: anteroposterior and mediolateral excursion of the center of pressure, speed of displacement of the center of pressure, length of postural ball and distribution of plantar pressures;
2. gait: spatio-temporal parameters, kinematics of trunk and joints of lower limbs, ground reaction forces, moments and joint powers.

A functional evaluation of the foot will be also performed positioning the patient prone/supine on the bed and measuring several joint angles.

The measurement will be supported by a video from which images can be subsequently processed to trace and obtain the joint angles.

For the functional evaluation of the hand, the patient will be evaluated with the following outcome measures:

1. Algo-functional index of the hand according to Dreiser, which analyzes the ability to execute some gestures of daily life;
2. Duruöz index, questionnaire for assessing functional impairment of hand.

ELIGIBILITY:
Inclusion Criteria:

* De novo patients with acromegaly (group # 1), diagnosed according to Endocrine Society guidelines,
* Age equal to18 years or older
* Acromegalic patients with different disease status (group #2)
* Age equal to18 years or older

Exclusion Criteria:

* Cardiorespiratory, neurological or musculoskeletal disorder
* Previous orthopaedic surgery
* Previous lower limbs traumatic injuries

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group #1: De novo patients with acromegaly, diagnosed according to Endocrine Society guidelines, aged equal or above 18 years old;
  Group #2: Acromegalic patients with different disease status (active disease despite ongoing therapies, controlled disease under medical therapy, and disease remission), aged equal or above 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-06-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in serum concentration of GH and IGF1 | At baseline in population #1 and # 2 and at 3, 6, 12 months after intervention in population #1
  Serum concentration of GH and IGF1
Change in postural | At baseline in population #1 and # 2 and at 3, 6, 12 months after intervention in population #1
  The postural evaluation was performed for 60 seconds while the participants were standing on a baropodometric platform (P-Walk, BTSBioengineering, Italy). They were instructed to maintain an upright position, with their eyes focused on a 6 cm black circle placed at their individual eye level, at a distance of 1.5 meters. Subsequently, they were asked to repeat the same task with their eyes closed. To avoid any learning or fatigue effects, two evaluations were acquired with open eyes and two with closed eyes, and between each trial, the subjects were allowed to rest and sit for 2 minutes, maintaining the foot position during the tests.
  Postural parameters were calculated using dedicated software (G-Studio, BTS, Italy). The relative range of the center of pressure track length is essentially the difference between the maximum and minimum CoP position in the anterior-posterior and medial-lateral (ML) directions during the maintenance of the upright posture.
Gait analysis | At baseline in population #1 and # 2 and at 3, 6, 12 months after intervention in population #1
  All participants were evaluated with 3D-Gait Analysis using an optoelectronic system composed of eight cameras (SMARTDX, BTSBioengineering, Italy) set at 100 Hz, and two force platforms (AMTI, USA). To evaluate the kinematics of each body segment, passive markers were positioned on the participants' body, as described by Davis III et al., and the underlying skeletal model was scaled on behalf of anthropometric data (height, weight, tibial length, distance between the femoral condyles or diameter of the knee, distance between the malleoli or diameter of the ankle, distance between the anterior iliac spines and thickness of the pelvis).
  After placing the markers, the participants were asked to walk barefoot at self-selected speed along a walkway where the force platforms were embedded. Kinematic and kinetic data were collected for each individual from at least five trials to guarantee the reproducibility of the results.
Change in function of the foot - angle ankle joint | At baseline in population #1 and # 2 and at 3, 6, 12 months after intervention in population #1
  The functional evaluation of the foot involves positioning the patient prone/supine on the bed and assessing the ankle joint
Change in function of the foot - angle subtalar joint | At baseline in population #1 and # 2 and at 3, 6, 12 months after intervention in population #1
  The functional evaluation of the foot involves positioning the patient prone/supine on the bed and assessing the subtalar joint
Change in function of the foot - angle metatarsophalangeal joint of the big toe | At baseline in population #1 and # 2 and at 3, 6, 12 months after intervention in population #1
  The functional evaluation of the foot involves positioning the patient prone/supine on the bed and assessing the metatarsophalangeal joint of the big toe
Change in Function of the hand - Dreiser functional index | At baseline in population #1 and # 2 and at 3, 6, 12 months after intervention in population #1
  Algo-functional index of the hand according to Dreiser functional index
Change in Function of the hand - Duruöz hand index | At baseline in population #1 and # 2 and at 3, 6, 12 months after intervention in population #1
  Algo-functional index of the hand according to Duruöz hand index

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Vitale, Principal Investigator — Istituto Auxologico Italiano IRCCS
Locations (1):
- Istituto Auxologico Italiano IRCCS San Luca, Milan, Italy